CLINICAL TRIAL: NCT06989827
Title: Evaluation of the Influence of Dry Eye Disease on the Precision of Preoperative Keratometry Measurements and Its Effect on Intraocular Lens Power Calculations in Patients Undergoing Cataract Surgery.
Brief Title: Impact of DED on the Accuracy of Preoperative Keratometry Values in the Calculation of IOL Power for Cataract Surgery.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Stjepan Pinotić, Medical Doctor, ophthalmology resident, University Hospital Sestre Milosrdnice
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DED_Cataract_25
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye Disease (DED); Cataract
Keywords: keratometry; IOL; intraocular lens; cataract surgery; dry eye disease; DED
MeSH Terms: conditions — Dry Eye Syndromes; Cataract

STUDY DESIGN:
Intervention Model Description: The study is designed to compare two parallel groups of patients, healthy controls and patients diagnosed with dry eye disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (No Intervention)
- Patients with diagnosed dry eye disease (Active Comparator)
  Interventions: Drug: Preservative free artificial tear

INTERVENTIONS:
Drug: Preservative free artificial tear — After diagnosing patients with dry eye disease we prescribed them preservative free artificial tears and scheduled them for a follow-up keratometry.
  Arms: Patients with diagnosed dry eye disease

SUMMARY:
This study looks at how dry eye disease can affect important eye measurements needed before cataract surgery. These measurements guide us in choosing the right artificial lens to implant, which is essential for achieving clear vision after the procedure. We are currently investigating whether patients with dry eyes tend to have less reliable readings due to surface irregularities on the eye. Our goal is to better understand this connection so we can improve pre-surgical preparation for patients with dry eye and help ensure better visual outcomes after cataract surgery.

DETAILED DESCRIPTION:
In this study, we are investigating the potential impact of dry eye disease (DED) on the accuracy of preoperative keratometry values used in intraocular lens (IOL) power calculations for cataract surgery. Precise keratometric measurements are essential for determining the appropriate IOL power to achieve optimal postoperative refractive outcomes. However, ocular surface irregularities associated with DED-such as tear film instability, corneal epithelial disruption, and increased surface variability-may compromise the repeatability and reliability of these measurements.

We aim to examine the correlation between the severity of dry eye and the variability or inaccuracy in keratometric readings obtained through standard biometry techniques. Patients undergoing cataract surgery are being prospectively evaluated and stratified based on dry eye status using established diagnostic criteria, including patient-reported symptom questionnaires (OSDI), tear break-up time (TBUT), corneal staining patterns (Oxford grading scale), Schirmer's test values, and Meibomian Gland Evaluation (Meibomian Quality Score). Preoperative keratometry data are collected using optical biometers, and repeated measurements are analyzed for variability. IOL power calculations are compared with postoperative refractive outcomes to assess clinical significance.

By identifying potential discrepancies linked to dry eye severity, we aim to determine whether preoperative DED management could meaningfully improve measurement precision and, consequently, visual outcomes. Preliminary observations suggest that untreated or suboptimally managed DED may lead to inconsistent keratometric values, which in turn could contribute to unexpected postoperative refractive errors.

Our ultimate goal is to provide evidence-based recommendations for preoperative screening and treatment protocols for DED in cataract surgery candidates. These findings could support the development of standardized guidelines that incorporate ocular surface optimization as an essential component of pre-surgical planning, thereby enhancing surgical precision and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls scheduled to undergo cataract surgery
* patients diagnosed with dry eye disease scheduled to undergo cataract surgery

Exclusion Criteria:

* patients already on therapy regimen using Preservative free artificial tears
* patients on antihistamines/decongestants, antidepressants, anti-Parkinson's, antipsychotics and antispasmodic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Variability in keratometric values before and after dry eye disease treatment with preservative free artificial tears | pre-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- UHC Sestre Milosrdnice, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang F, Yang L, Ning X, Liu J, Wang J. Effect of dry eye on the reliability of keratometry for cataract surgery planning. J Fr Ophtalmol. 2024 Feb;47(2):103999. doi: 10.1016/j.jfo.2023.04.016. Epub 2023 Oct 31. PMID 37919153